CLINICAL TRIAL: NCT06400628
Title: Effectiveness of Chronic Self-management Education on Behavioral and Clinical Outcomes of Patients With Rheumatic Heart Disease at Jimma Medical Center (JMC): A Pseudo Quasi Experimental Design
Brief Title: Effectiveness of Chronic Self-management Education on Behavioral and Clinical Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jimma University (Other)
Responsible Party: Principal Investigator, Hiwot Berhanu, Assistant professor, Jimma University
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: JUIH/IRB/277/23.
Record Dates: First submitted 2024-04-15; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Rheumatic Fever; Rheumatic Diseases
MeSH Terms: conditions — Rheumatic Fever; Rheumatic Diseases

STUDY DESIGN:
Intervention Model Description: Participants will be randomly selected to be included in the study. Once included, baseline data will be collected from the participants on the date of inclusion, which will serve as the control group or Arm 1 data. Subsequently, all participants will receive an educational intervention, consisting of one-to-one nurse-led multi-component chronic disease self-management education (CDSME), for four consecutive months. During this time, the indicated variables, including blood pressure, pulse rate, weight, and complete blood count, will be measured during monthly visits. Finally, the same variables of the base line variables will be measured from the participants and serve as the second arm (arm2). The study aims to recruit 166 patients with rheumatic heart disease (RHD) from the Jimma Medical Center cardiac clinic.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: participants and investigator were informed about the expected outcomes. However, care providers and outcome assessor were masked to overcome any associated bias
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- initial and end (Active Comparator)
  Interventions: Behavioral: Self-management education
- Quasi experimental design (Experimental): quasi
  Interventions: Behavioral: Self-management education

INTERVENTIONS:
Behavioral: Self-management education — The base line data will be taken and used as control, while the final result will be utilized as the case

SUMMARY:
Study Design, Setting, and Period A one-group quasi-experimental study using a pre-test and post-test will be implemented on a convenient sample design to examine the effectiveness of chronic disease self-management education in improving clinical outcomes and decreasing depression and anxiety among patients under medical follow-up at Jimma Medical Center cardiac clinic.

A comprehensive evaluation of both clinical and laboratory measurements will be conducted before and after the education intervention. Education will be provided monthly, four times (at 30, 60, 90, and 120 days), with data collection occurring over four months.

Sample Size, Sampling Technique, and Criteria The participants in this study will be patients diagnosed with rheumatic heart disease at Jimma Medical Center cardiac clinic who visit the outpatient department for medical follow-up. The study will introduce multi-component nurse-led chronic disease self-management education interventions. It will involve a pretest followed by an educational session and a post-test conducted with a one-to-one face-to-face education section. The duration of each session will vary between 30 and 45 minutes based on the participants' needs.

The sample size for the study will be determined using Rao software, considering parameters such as a margin of error of 5%, a confidence level of 95%, a monthly population size of 315, and an unknown response distribution with a conservative estimate of 50%. Based on these factors, the calculated sample size will be 174 study subjects.

Data Analysis Data analysis will be conducted using Statistical Package for the Social Sciences (SPSS) version 25.0. Values will be presented as mean ± standard deviation (SD) for continuous variables and percentage for categorical variables. Continuous data will be compared using a two-tailed Student t-test. A p-value of less than 0.05 will be considered statistically significant for all tests conducted.

DETAILED DESCRIPTION:
Measurements In this study, blood samples will be collected from participants using the syringe technique, and the samples will be analyzed using a five-differential cellular analysis system machine manufactured by Beckman Coulter in Ireland. The machine will generate flags indicating certain abnormalities in the blood parameters. To confirm these flags and assess the performance of the automated hematology analyzer, a peripheral blood morphology examination will be conducted. For this examination, a thin blood smear will be prepared from the CBC sample, air-dried, and then stained with Wright stain. Laboratory technologists will carefully examine the stained smear using a 100X oil immersion objective to assess the morphology of red blood cells.

To evaluate anxiety and depressive symptoms among patients with rheumatic heart disease (RHD), the participants will be provided with the Amharic version of the Hospital Anxiety and Depression Scale (HADS). This scale consists of 14 items, which are divided into two subscales: one for depression and the other for anxiety. Each item on the scale is scored from 0 to 3, with 0 representing the lowest severity and 3 indicating the highest severity of anxiety or depression. The scores on the subscales will be summed up to obtain a final score, ranging from 0 to 21. Based on the score counts, three levels will be established: normal (0-7), borderline (8-10), and abnormal (11-21). These levels provide guidance for assessing the severity of anxiety and depression symptoms in the participants.

Weight and height will be measured using a combined height and weight scale (made in India, manufactured on March 17, 2017). Weight will be measured to the nearest 0.1 kg with the participant not wearing shoes and heavy clothes, whereas height will be measured to the nearest 0.1 cm with the participant standing upright with the heel, buttock, and upper back along the same vertical plane, arms at the side, and looking straight forward. Blood pressure will be measured on the left arm in mmHg using a calibrated sphygmomanometer (Yton sphygmomanometer, Italy, model 10220060) while the participant is in a sitting position with his/her back supported, legs uncrossed, arm supported, and cubital fossa at heart level after 5 minutes of resting arms at the side and looking straight forward.

Tools and protocols for chronic disease self-management education The self-management education program includes information about the structure and function of the heart, disease risk factors, symptoms management, prophylaxis (penicillin/oral antibiotics) and/or medication compliance, nutrition and dietary management, as well as maintaining a healthy daily lifestyle. The education session will be developed based on heart failure management guidelines produced by the American Heart Failure Society, the Joanna Briggs Institute's (JBI) evidence-based manual, and the Ethiopian Ministry of Health. All the patients to be enrolled in a series of educational sessions will be led by experienced nurse educators.

The contents of the program will be reviewed by experts in cardiology, nutrition, and public health. Face-to-face education methods will be established, and the participants will be provided with an educational leaflet with information about RHD, heart failure, self-reported symptoms, and self-care behavior.

1. Understanding rheumatic heart disease and self-management of heart failure 1. Introduction Education 2. Knowledge about RHD and heart failure Definition, etiology, symptoms, complications, diagnosis, and treatment 3. Updating the patient's current disease status Medications, complications 4. Self-management of heart failure in patients with RHD

   - Management of symptoms, medication, nutrition, emotions, and daily life
2. Symptoms Monitor the symptoms of patients on a monthly basis and during their unscheduled follow-up visits.

   * Assess the factors that worsen and alleviate the symptoms. 2. Verify the use of self-symptom checklists and self-care behavior calendar.
   * Evaluate and implement strategies for managing and retraining Education

     1. Symptoms of heart failure, measure
     2. Signs of heart failure requiring immediate attention, assessment
     3. Discussion, question, and answer
3. Prophylaxis and medication Education 1. Importance of Prophylaxis in preventing the recurrence of Acute rheumatic fever and disease severity

   * Schedule regular follow-up visits, Injection site care Common side effect of benzathine penicillin 2. Types of medication, effects, and side effects 3. Side effects and toxicity of the drug of heart failure 4. Providing information about the medication's details and purpose. 5. Assessing the challenges and potential adverse reactions associated with the medication/prophylaxis.

     6. Establish a routine follow-up for consistent medication and prophylaxis usage through the utilization of a self-care behaviors calendar 7. Question and answer 4. Nutrition

     1. Education
   * Dietary considerations for individuals with heart failure.
   * Restrictions on dietary intake of salt, fluid
   * Importance of a balanced diet and meal plan
   * Important dietary factors to consider for individuals taking warfarin medication.
   * Develop a routine of regularly monitoring weight as frequently as possible.
   * Question and answer 5.Routine, daily living Education Relaxation, stress management, Avoid alcohol intake, khat chewing, and smoking Incorporate a regular physical activity routine by utilizing a self-care behaviors calendar.

Question and answer

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria

* Patients aged 15 years and above with verified diagnosis through echocardiography imaging.
* Patients diagnosed as rheumatic heart disease for at least 6 months by a cardiologist. New York Heart Association (NYHA) function Class II/III.
* Participants who possess the ability to effectively communicate, comprehend the study objectives, and
* Provided consent to participate in the research.

Exclusion Criteria:

* Patients under serious medical conditions,
* The existence of chronic illnesses like chronic obstructive pulmonary disease or asthma, diabetes, chronic kidney failure, stroke, or advanced-stage cancer.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Pre- and post-systolic blood pressure, diastolic blood pressure | Four for months
  The effectiveness of the study will be assessed through the measurement of pre and post blood pressure. Blood pressure will be measured using a sphygmomanometer
pre and post weight measurements | Four four months
  weight will be measured using a combined height and weight scale.
Pre- and post- anxiety and depression levels | Four four months
  Pre- and post- anxiety and depression levels using the Hospital Anxiety and Depression scale Questionnaire (HADS)
Pre and post complete blood count | Four four months
  automated hematology analyzer will be used to quantities cells in a person's blood.

CONTACTS AND LOCATIONS:
Locations (1):
- Jimma university, Jimma, Oromi, Ethiopia

IPD SHARING:
Plan to Share IPD: No
Clinical and RHD indicting laboratory parametric measurements will be measured at initial stage and compared with final measurement results